CLINICAL TRIAL: NCT05762705
Title: A Multisite Randomized Trial of Viral Combat: A Mobile Gaming App to Improve Adherence to PrEP
Brief Title: A Mobile Gaming App to Improve Adherence to PrEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00067477
Record Dates: First submitted 2023-02-12; First posted 2023-03-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Medication Adherence; HIV/AIDS
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multilevel Gaming Adherence (Experimental): Participants in the intervention arm will receive Multilevel Gaming Adherence Intervention. Participants receive Viral Combat on their mobile phones, and, for 24 weeks, game-related text messages guided by self-reported medication adherence.
  Interventions: Behavioral: Multilevel Gaming Adherence Intervention
- Treatment as Usual + (Active Comparator): TAU+ participants will receive the Treatment As Usual + intervention, which includes receiving a non-HIV related mobile game.
  Interventions: Behavioral: Treatment as Usual +

INTERVENTIONS:
Behavioral: Multilevel Gaming Adherence Intervention — Information-Motivation-Behavior based mobile gaming application tailored for those taking PrEP and adherence-based text messages
  Arms: Multilevel Gaming Adherence
Behavioral: Treatment as Usual + — non-PrEP related mobile gaming application
  Arms: Treatment as Usual +

SUMMARY:
In this study, the investigators will test the mobile game, Viral Combat, for efficacy and acceptability among diverse participants, ages 15-34 years, receiving PrEP care in clinical settings in New England and Mississippi. Formative evaluation interviews will be conducted with stakeholders (healthcare workers, clinic administrators, and patients taking PrEP) to inform intervention delivery. Data from the formative interviews will also be used to make necessary adaptations to the game and assess acceptability for diverse populations and clinics. Viral Combat will then be further tested with 200 participants ages 15-34 years, receiving PrEP care at clinical sites in the South (n=100 Jackson, MS) and New England (n=100, Providence, RI; Boston, MA) in a multisite Hybrid Type 1 effectiveness-implementation randomized controlled trial (RCT). This trial will test the efficacy of the intervention compared to a control condition (a non-PrEP related game) on biological and behavioral measures. At the end of the trial, a summative evaluation of the implementation context using the i-PARIHS framework will occur. These interviews with study participants and clinic staff will inform future implementation and dissemination of Viral Combat.

DETAILED DESCRIPTION:
In this study, the investigators will test the mobile game, Viral Combat, for efficacy and acceptability among diverse participants, ages 15-34 years, receiving PrEP care in clinical settings in New England and Mississippi. Formative evaluation interviews will be conducted with stakeholders (healthcare workers, clinic administrators, and patients taking PrEP) to inform intervention delivery. Data from the formative interviews will also be used to make necessary adaptations to the game and assess acceptability for diverse populations and clinics. Viral Combat will then be further tested with 200 participants ages 15-34 years, receiving PrEP care at clinical sites in the South (n=100 Jackson, MS) and New England (n=100, Providence, RI; Boston, MA) in a multisite Hybrid Type 1 effectiveness-implementation randomized controlled trial (RCT). This trial will test the efficacy of the intervention compared to a control condition (a non-PrEP related game) on biological and behavioral measures. At the end of the trial, a summative evaluation of the implementation context using the i-PARIHS framework will occur. These interviews with study participants and clinic staff will inform future implementation and dissemination of Viral Combat.

Aim 1: To conduct formative evaluation interviews, guided by the i-PARHIS framework, with approximately 30 stakeholders (23 PrEP patients, 4 clinical staff, 3 clinic administrators) in order to adapt Viral Combat for diverse PrEP patient populations, and to identify individual, organizational, and structural factors associated with its implementation.

Aim 2: To evaluate, in a Hybrid Type 1 effectiveness-implementation randomized controlled trial with 200 participants taking PrEP (15-34 years of age), the effectiveness of Viral Combat compared to a control group that receives a non-PrEP related game.

The investigators will examine the impact of the intervention on:

2a: improving adherence to PrEP using a biological measure (tenofovir from DBS), clinic records, and self-report; 2b: the potential mediators of the intervention, such as knowledge, motivation, self-efficacy, and game metrics.

Aim 3: To conduct summative evaluation interviews, following the RCT phase, with an additional 30 stakeholders ((23 PrEP patients, 4 clinical staff, 3 clinic administrators). Interviews will assess and summarize the i-PARIHS constructs relevant to the intervention's future implementation success.

ELIGIBILITY:
Inclusion Criteria:

* 15-34 years old
* English speaking
* Initiated PrEP in the last 30 days or re-initiated PrEP after not taking PrEP for at least 1 month
* HIV negative as per clinician and clinical record
* Able to give consent/assent and not impaired by cognitive or medical limitations as per clinical assessment.

Exclusion Criteria:

* None

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Tenofovir (TFV) blood concentration at 24 weeks | 24 weeks
  Tenofovir (TFV) concentration in blood from either venipuncture or dried blood spot labs immediately post-intervention (at 24 weeks follow-up).

SECONDARY OUTCOMES:
Tenofovir (TFV) blood concentration at 48 weeks | 48 weeks
  Tenofovir (TFV) concentration in blood from either venipuncture or dried blood spot labs at the end of study follow-up (at 48 weeks follow-up).
Self-reported Medication Adherence at 24 weeks | 24 weeks
  Proportion of days with missed doses via self-report: (reported missed doses in past month) / (total number of days in month) immediately post-intervention (at 24 weeks follow-up).
Self-reported Medication Adherence at 48 weeks | 48 weeks
  Proportion of days with missed doses via self-report: (reported missed doses in past month) / (total number of days in month) at the end of study follow-up (at 48 weeks follow-up).
Medical appointment adherence at 24 weeks | 24 weeks
  Number of PrEP-related medical visits kept in the past 3 months based on clinic records at 24 weeks follow-up.
Medical appointment adherence at 48 weeks | 48 weeks
  Number of PrEP-related medical visits kept in the past 3 months based on clinic records at 48 weeks follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brock, MD, Study Director — Rhode Island Hospital; Sharon Vuppula, MD, Study Director — Boston Medical Center
Locations (3):
- United States (3):
  - Boston Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Lifespan (The Miriam Hospital and Rhode Island Hospital), Providence, Rhode Island